CLINICAL TRIAL: NCT00114439
Title: An Open Label Trial of Lithium for the Management of Cannabis Withdrawal
Brief Title: Lithium Cannabis Withdrawal Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sydney South West Area Health Service (Other Government)
Collaborators: The University of New South Wales (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSWAHS HREC 2005/047; UNSW HREC 04168
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Cannabis Dependence; Substance Withdrawal Syndrome
Keywords: cannabis withdrawal; lithium; Cannabis withdrawal syndrome
MeSH Terms: conditions — Marijuana Abuse; Substance Withdrawal Syndrome | interventions — Lithium Carbonate

INTERVENTIONS:
Drug: Lithium carbonate

SUMMARY:
This trial will examine the efficacy of lithium in providing symptomatic relief from the withdrawal discomfort experienced by some dependent users of cannabis on cessation of regular use. Significant withdrawal may be a barrier to achieving abstinence in some clients and can be associated with marked disturbances in mood, sleep, hostility and aggression. Relief from such symptoms may be important in helping some clients achieve a period of abstinence and facilitate subsequent entry into a relapse prevention program.

DETAILED DESCRIPTION:
There are currently no accepted pharmacotherapies for the management of cannabis withdrawal. A recent study by Cui et al (2001) investigated the effects and mechanism of lithium on cannabinoid withdrawal in rats. The researchers found that lithium administration prevented the development of withdrawal symptoms, and suggested that increased oxytocin secretion resulting from lithium dosing prevented the withdrawal syndrome from occurring. Although caution should be exercised in generalising the results of an animal study, preliminary results of a small pilot study in humans are consistent with the potential utility of lithium in the management of human cannabis withdrawal (Zhang, personal communication). Furthermore, human use of lithium is well established and the addition of a readily available drug such as lithium carbonate would be a useful clinical tool should it prove efficacious in a series of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of cannabis dependence with at least a three-month history.
* Seeking treatment for primary cannabis problem
* Withdrawal identified as barrier to abstinence

Exclusion Criteria:

* Other drug dependency (excluding nicotine)
* Client is breastfeeding or pregnant.
* Client has contraindicated medical or psychiatric conditions.
* Client currently taking other medications that may interact with lithium.
* Known hypersensitivity / side effects with Lithium.
* Currently receiving Lithium from another source.
* Currently prescribed any antidepressant / mood stabilising / antipsychotic medication.
* Currently receiving opioid pharmacotherapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2005-09; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Severity of reported cannabis withdrawal symptoms
Treatment retention
Cannabis use
Depression
Anxiety
Aggression/Anger
Sleep difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Adam R Winstock, MBBS BSc MSc MRCP(UK) MRCP, Principal Investigator — Corella Drug Treatment Service
Locations (1):
- Corella Drug Treatment Service, Fairfield, New South Wales, Australia

REFERENCES:
- [Background] Cui SS, Bowen RC, Gu GB, Hannesson DK, Yu PH, Zhang X. Prevention of cannabinoid withdrawal syndrome by lithium: involvement of oxytocinergic neuronal activation. J Neurosci. 2001 Dec 15;21(24):9867-76. doi: 10.1523/JNEUROSCI.21-24-09867.2001. PMID 11739594